CLINICAL TRIAL: NCT01857427
Title: A Prospective Observational Cohort to Study the Genetics of Obstructive Sleep Apnea and Associated Co-Morbidities
Status: Active, not recruiting | Type: Observational
Sponsor: Ulysses Magalang MD (Other)
Responsible Party: Sponsor-Investigator, Ulysses Magalang MD, Professor of Internal Medicine, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0214
Record Dates: First submitted 2013-05-10; First posted 2013-05-20 (Estimated); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood or saliva sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The primary objective of this study is to build a well characterized cohort of patients that will be used to determine the genetic variants associated with obstructive sleep apnea (OSA)and its co-morbidities.

DETAILED DESCRIPTION:
The purpose of building the cohort is to allow the performance of genome-wide association studies with a large sample of patients that have been well-characterized using standardized procedures.

ELIGIBILITY:
Inclusion Criteria:

We will recruit subjects who are:

* 18 years of age and older.
* Willing and able to give informed consent

AND any of the following:

* PSG (polysomnogram)requested by a physician based on clinical grounds
* AHI (Apnea-hypopnea index) ≥ 5 episodes per hour based on a prior PSG.

Exclusion Criteria:

Incapable of giving informed consent

* Under the age of 18

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects 18 years of age and older who are scheduled for polysomnography (PSG), regardless of final diagnosis AND adult subjects who have already been diagnosed with OSA based on a prior PSG and are already on treatment. OSA diagnosis will be defined as an apnea/hypopnea index (AHI) >or =5 episodes per hour.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sleep Questionnaire | upon enrollment
  Responses to sleep questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- Suite 2600, Martha Morehouse Medical Pavilion, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No